CLINICAL TRIAL: NCT01630018
Title: A Phase Ⅱb, Randomized, Open, Parallel-Group, Multi-Center Trial to Assess the Efficacy and Safety of Belotecan(CamtoBell Inj.) or Topotecan in Patients With Recurrent or Refractory Ovarian Cancer
Brief Title: Belotecan Versus Topotecan for Recurrent Ovarian Cancer: A Randomized, Open-label, Parallel-group Phase IIb Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11AOC09J
Record Dates: First submitted 2012-03-06; First posted 2012-06-28 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Belotecan; Topotecan
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Topotecan; belotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topotecan (Active Comparator): Topotecan
  Interventions: Drug: Topotecan
- Camtobell (Active Comparator): Belotecan
  Interventions: Drug: Belotecan

INTERVENTIONS:
Drug: Topotecan — 1.5mg/m2 IV days 1,2,3,4,5 of each 21day cycle until 6cycle or disease progression
  Other Names: Hycamtin inj.
  Arms: Topotecan
Drug: Belotecan — 0.5mg/m2 IV days 1,2,3,4,5 of each 21day cycle until 6cycle or disease progression
  Other Names: Camtobell inj.
  Arms: Camtobell

SUMMARY:
The purpose of this study is to determine the efficacy and safety of belotecan or topotecan in patients with recurrent or refractory ovarian cancer (AOC).

DETAILED DESCRIPTION:
A Phase Ⅱb, Randomized, Open, Parallel-Group, Multi-Center Trial to Assess the Efficacy and Safety of Belotecan (CamtoBell inj.) or Topotecan in Patients with Recurrent or Refractory Ovarian Cancer

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histological or cytological diagnosis of AOC
* Stable disease (SD) or progression at time of study entry Recurrent or progressive AOC ≥ 90 days of duration of response for first-line therapy
* Measurable disease defined by RECIST criteria
* ECOG Performance Status of 0, 1, or 2
* Life expectancy > 3 months
* Adequate bone marrow, Renal, Hepatic reserve:

  * absolute neutrophil (segmented and bands) count (ANC) ≥ 1500 cells/μL
  * platelet count ≥ 100,000 cells/μL
  * hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 X ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 X ULN
  * Alkaline Phosphatase (ALP) ≤ 2.0 X ULN
  * Serum creatinine < 1.5mg/dL or calculated creatinine clearance > 60mL/min
* Signed a written informed consent

Exclusion Criteria:

* Active infection
* Symptomatic brain lesion
* Any other type of cancer during the previous 5 years except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix Severe concurrent diseases
* Prior anticancer therapy within 4 weeks before enroll
* Active pregnancy test and Pregnant or nursing women
* Participation in any investigational drug study within 28 days prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate | approximately 21 days(every 1 Cycle)

SECONDARY OUTCOMES:
Overall Survival | up to 4 years
Progression Free survival | up tp 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Sang Song, phD, Dr, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul Metropolitan, South Korea

REFERENCES:
- [Derived] Kim HS, Park SY, Park CY, Kim YT, Kim BJ, Song YJ, Kim BG, Kim YB, Cho CH, Kim JH, Song YS. A multicentre, randomised, open-label, parallel-group Phase 2b study of belotecan versus topotecan for recurrent ovarian cancer. Br J Cancer. 2021 Jan;124(2):375-382. doi: 10.1038/s41416-020-01098-8. Epub 2020 Sep 30. PMID 32994466